CLINICAL TRIAL: NCT03196518
Title: PET Imaging of Thyroid Tissue Expressing Sodium-iodine Symporter Using the New Tracer 18F-tetrafluoroborate (18F-TFB)
Brief Title: Study of PET Imaging With 18F-TFB in Patients With Thyroid Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-315
Record Dates: First submitted 2017-06-21; First posted 2017-06-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Cancer
Keywords: PET Imaging; 18F-TFB; 17-315
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: This is a pilot study evaluating the safety, radiation dosimetry and detection capability of 18F-tetrafluoroborate (18F-TFB), a novel tracer for sodium-iodine symporter (NIS) imaging.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET Imaging With 18F-TFB (Experimental): The intervention is the administration of a single dose of approximately 5-10 mCi 18F-TFB (mass <= 50 μg) for imaging purposes. This will be followed by a 30 minute dynamic PET/CT study immediately after injection, at 60 minutes (+/- 10 min) and 4 hours (+/- 15 min) post injection. The second and third scan will last up to 30 minutes.
  Interventions: Procedure: PET Imaging; Other: 18F-tetrafluoroborate (18F-TFB)

INTERVENTIONS:
Procedure: PET Imaging — PET/CT study immediately after injection
Other: 18F-tetrafluoroborate (18F-TFB) — administration of a single dose of approximately 5-10 mCi 18F-TFB (mass <= 50 μg) for imaging purposes

SUMMARY:
The goal of the study is to evaluate a new imaging test that may allows the investigators to predict the uptake of radioactive iodine by thyroid cancer faster than the current standard and that does not interfere with the uptake of radioactive iodine used for therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed thyroid carcinoma of follicular origin (including papillary and its respective variants).
* Patients should have tumors that are radiographically evident on PET, ultrasound, CT or MRI
* Age ≥ 18 years.
* ECOG performance status ≤ 2 (or Karnofsky ≥60%).
* Patients must have normal organ and bone marrow function as defined below:

  * Absolute neutrophil count (ANC) > 1.5x10^9/L
  * Hemoglobin ≥ 9 g/dL
  * Platelets ≥ 100 x 10^9/L
  * Albumin ≥ 2.5 g/dL
  * Total bilirubin ≤ 1.5x institutional ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2x institutional ULN unless it is related to the primary disease
  * Creatinine ≤ 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) ≥ 50 mL/min OR 24-hour urine creatinine clearance ≥ 50 mL/min
* Negative pregnancy test within 7 days prior to starting the study in premenopausal women. Women of non-childbearing potential may be included without pregnancy test if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
* Fertile men and women must use an effective method of contraception during treatment and for at least 6 months after completion of treatment as directed by their physician. Effective methods of contraception are defined as those, which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (for example implants, injectables, combined oral contraception or intra-uterine devices). At the discretion of the Investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant, lactating, or breast feeding women.
* Patients unable to follow a low iodine diet or requiring medication with high content in iodide (amiodarone).
* Patients who received iodinated intravenous contrast as part of a radiographic procedure within 3 months of study registration. Those that have had iodinated intravenous contrast for CT imaging within this time frame may still be eligible if a urinary iodine analysis reveals that the excess iodine has been adequately cleared after the last intravenous contrast administration.
* Unwillingness or inability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety Outcome Measures (CTCAE v4) severity of adverse events | up to 2 day following scan
  Safety Outcome Measures (CTCAE v4) severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Grewal, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Backhaus P, Pentlow KS, Ho AL, Mauguen A, Fagin JA, Pillarsetty NVK, Lyashchenko SK, Burnazi E, Ghossein RA, Chhabra S, Abusamra M, Larson SM, Schoder H, O'Donoghue J, Weber W, Grewal RK. [18F]TFB PET/CT misses intense [124I]iodine-avid metastases after redifferentiation therapy in metastatic thyroid cancer. EJNMMI Res. 2024 Oct 8;14(1):91. doi: 10.1186/s13550-024-01138-x. PMID 39377970
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm